CLINICAL TRIAL: NCT00052715
Title: Phase II Trial Of Poly-ICLC For Glioblastoma
Brief Title: Biological Therapy and Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Acronym: Poly-ICLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: prematurely discontinued after results of the EORTC phase-3 study defined the SOC for newly diagnosed GMB pts as RT plus concomitant and adjuvant TMZ
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NABTC-0105; CDR0000258685 (Registry Identifier: PDQ (Physician Data Query)); NCI-2012-02506 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- poly-ICLC Newly diagnosed GBM (Experimental): Poly-ICLC 20ug/kg 3 times a week (Monday-Wednesday-Friday) starting one week before Radiation Therapy
  Intramuscular injection
  Drug Poly-ICLC
  Interventions: Drug: poly ICLC

INTERVENTIONS:
Drug: poly ICLC

SUMMARY:
RATIONALE: Biological therapies such as poly-ICLC use different ways to stimulate the immune system and stop tumor cells from growing. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining biological therapy with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining poly-ICLC with radiation therapy in treating patients who have newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of poly ICLC and radiotherapy, in terms of total survival from date of diagnosis, in patients with newly diagnosed glioblastoma multiforme.
* Determine the safety and toxicity profile of this regimen in these patients.
* Determine the 12-month survival rate in patients treated with this regimen.
* Assess progression-free survival at 6 months and median progression-free survival from date of diagnosis of patients treated with this regimen.
* Assess response in patients treated with this regimen.
* Assess changes in neurological status in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Within 1-4 weeks after surgery, patients receive poly ICLC intramuscularly 3 times weekly (on days 1, 3, and 5). Treatment continues in the absence of disease progression or unacceptable toxicity.

One week after the initiation of poly ICLC, patients undergo external beam radiotherapy once daily 5 days a week for 6 weeks.

Patients are followed monthly for 1 year and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed intracranial glioblastoma multiforme (GBM) or gliosarcoma by biopsy or resection within the past 28 days

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* More than 8 weeks

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL (transfusion allowed)

Hepatic

* Bilirubin less than 2 times upper limit of normal (ULN)
* SGOT less than 2 times ULN

Renal

* Creatinine less than 1.5 mg/dL

Other

* No significant medical illness that cannot be controlled adequately with appropriate therapy or that would compromise tolerability of study therapy
* No other cancer (except nonmelanoma skin cancer or carcinoma in situ of the cervix) unless in complete remission and off all therapy for that disease for at least 3 years
* No active infection
* No disease that would obscure toxicity or dangerously alter drug metabolism
* No other serious concurrent medical illness
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior polifeprosan 20 with carmustine implant (Gliadel wafer)
* No concurrent chemotherapy

Endocrine therapy

* Concurrent corticosteroids to treat symptoms or prevent complications are allowed

Radiotherapy

* No prior radiotherapy to the brain
* No concurrent stereotactic radiosurgery
* No concurrent brachytherapy

Surgery

* See Disease Characteristics

Other

* No prior cytotoxic or noncytotoxic drug therapy for GBM
* No prior experimental drug therapy for GBM
* No other concurrent cytotoxic or noncytotoxic drug therapy for GBM
* Concurrent analgesics, antiepileptics, or other drugs to treat symptoms or prevent complications are allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2002-10-23 (Actual); Primary Completion 2006-02-25 (Actual); Study Completion 2009-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Prados, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Comprehensive Cancer Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Butowski N, Chang SM, Junck L, DeAngelis LM, Abrey L, Fink K, Cloughesy T, Lamborn KR, Salazar AM, Prados MD. A phase II clinical trial of poly-ICLC with radiation for adult patients with newly diagnosed supratentorial glioblastoma: a North American Brain Tumor Consortium (NABTC01-05). J Neurooncol. 2009 Jan;91(2):175-82. doi: 10.1007/s11060-008-9693-3. Epub 2008 Sep 17. PMID 18797818

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from 7/14/2003 through 12/19/2005. Patients recruited from outpatient clinic centers.
Groups:
- Poly-ICLC: poly-ICLC given at dose of 20mcg/kg 3 times weeekly by intramusclular injection. days of administration were at least 2 days apart. Mon-Wed-fri
  Poly-ICLC drug
  poly ICLC
Period: Overall Study
Arm/Group | Poly-ICLC
Started | 31
Completed | 30
Not Completed | 1
Not completed — wrong histology | 1

BASELINE CHARACTERISTICS:
Arm/Group | Poly-ICLC
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 53 [26 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 0
  Unknown or Not Reported | 1
Karnofsky Performance Status Scale [Median (Full Range); unit: units on a scale] — Higher score better 100 normal no complaints/disease 90 capable normal activity few symptoms/disease 80 normal activity, some difficulty some symptoms/signs 70 caring for self not capable normal activity/work 60 requiring some help can take care of most personal requirements 50 requires help often requires frequent medical care 40 disabled requires special care/help 30 severely disabled hospital admission indicated but no risk of death 20 very ill urgently requiring admission requires supportive measures/treatment 10 moribund rapidly progressive fatal disease processes 0 death
  units on a scale | 90 [60 to 100]
Histology Glioblastoma [Number; unit: participants] — WHO Classification
  participants | 30
Extent of Resection [Count of Participants; unit: Participants]
  Biopsy | 2
  Subtotal resection | 17
  Gross Total resection | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival in Pts With Newly Diagnosed GBM
Description: Overall survival from surgical diagnosis in patients with Newly Diagnosed GBM
Time Frame: 2 years
Population: Four patents were censored for survival at 35, 114, 126, and 166 weeks
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Poly-ICLC Newly Diagnosed GBM: Poly-ICLC 20ug/kg 3 times a week (Monday-Wednesday-Friday) starting one week before Radiation Therapy
  Intramuscular injection
  Drug Poly-ICLC
  poly ICLC
Arm/Group | Poly-ICLC Newly Diagnosed GBM
Number analyzed (Participants) | 30
weeks | 65 [54.8 to 74.2]

2. Secondary Outcome: To Determine 6 Months Progression Free Survival
Description: Patients evaluated from date of diagnosis to the 6 month scan
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Poly-ICLC Newly Diagnosed GBM
Number analyzed (Participants) | 30
percentage of participants | 30

3. Secondary Outcome: Determine the 12-month Survival Rate
Description: 12-month survival rate calculated from date of diagnosis
Time Frame: 1 year
Measure: Number; unit: percent of participants
Arm/Group | Poly-ICLC Newly Diagnosed GBM
Number analyzed (Participants) | 30
percent of participants | 69

4. Secondary Outcome: to Determine Grade 3 and 4 Toxicities Associated With Poly-ICLC in Newly Diagnosed Patients
Description: CTCAE 4
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Poly-ICLC Newly Diagnosed GBM
Number analyzed (Participants) | 30
participants
  Fatigue | 4
  Leukopenia | 4
  Lymphocytopenia | 2
  Myalgia | 1
  Fever without infection | 1
  Thrombosis | 2
  Pain | 1
  Rigor/Chills | 1

5. Secondary Outcome: To Determine the Change in Neurological Status in Patients With Glioblastoma Treated With External Beam Radiotherapy and Poly-ICLC
Description: Descriptive measure per investigator to describe change in neurological status post-intervention.
Time Frame: 1 year
Population: Data was not collected for this outcome measure due to premature discontinuation of study agent in response to what turned out to be pseudo-progression.
Arm/Group | Poly-ICLC Newly Diagnosed GBM
Number analyzed (Participants) | 0

6. Secondary Outcome: To Determine Tumor Response
Description: Tumor response to treatment with Poly-ICLC
Time Frame: 2 years
Population: Data was not collected for this outcome measure due to reports of transient enlargement of contrast enhancing disease with subsequent shrinkage during Poly-ICLC treatment and the lack of central radiological review, the protocol defined criteria for radiological response could not be employed because of the risk of inconsistent results
Arm/Group | Poly-ICLC Newly Diagnosed GBM
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Poly-ICLC
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 30/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Poly-ICLC (N=30)
Fatigue (General disorders) | 24 (24)
Pain (Other) (Musculoskeletal and connective tissue disorders) | 11 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (10)
Lymphocytopenia (Blood and lymphatic system disorders) | 9 (9)
Rigors/chills (General disorders) | 9 (9)
Alanine Aminotransferase Increased (Investigations) | 7 (7)
Granulocytopenia (Blood and lymphatic system disorders) | 7 (7)
Alkaline Phosphatase Increased (Investigations) | 6 (6)
Aspartate Aminotransferase Increased (Investigations) | 6 (6)
Headache (Nervous system disorders) | 6 (6)
nausea (Gastrointestinal disorders) | 5 (5)
alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Anorexia (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Fever (General disorders) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 4 (4)
Weight Loss (Gastrointestinal disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Blood Bilirubin Increase (Investigations) | 2 (2)
Hyperidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Gastrointestinal Other (Gastrointestinal disorders) | 2 (2)
Infection Other (Infections and infestations) | 2 (2)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Seizure (Nervous system disorders) | 2 (2)
Neuropathy Sensory (Nervous system disorders) | 2 (2)
Speech Impairment (Nervous system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Enrollment was prematurely discontinued after the results of the EORTC phase-3 study defined the standard of care for newly diagnosed glioblastoma patients as radiotherapy plus concomitant and adjuvant temozolomide (2005)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No